CLINICAL TRIAL: NCT01887119
Title: Effects of Aldosterone Antagonism on Insulin-mediated Microvascular Function in Subjects With the Metabolic Syndrome
Brief Title: Aldosterone Antagonism and Microvascular Function
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit sufficient participants
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Monica Schütten, MD, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 133031
Record Dates: First submitted 2013-06-19; First posted 2013-06-26 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Abdominal Obesity Metabolic Syndrome; Insulin Resistance; Hypertension
MeSH Terms: conditions — Abdominal obesity metabolic syndrome; Insulin Resistance; Hypertension | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eplerenone (Active Comparator): Eplerenone 50 mg 1dd during four weeks
  Interventions: Drug: Eplerenone
- Placebo (Placebo Comparator): Eplerenone-matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Eplerenone
  Arms: Eplerenone
Other: Placebo — Eplerenone-matched placebo
  Arms: Placebo

SUMMARY:
The prevalence of obesity and obesity-related complications is currently taking epidemic proportions. These complications increase the risk of type 2 diabetes and cardiovascular disease, which are important causes of morbidity and mortality worldwide.

It is important to gain insight in the mechanisms underlying obesity-related complications, because this may lead to the development of directed therapeutic strategies.

Currently, there is significant evidence that the cause of both insulin resistance and hypertension must be sought at the level of the microcirculation.

Over activity of the renin-angiotensin-aldosterone system is a potential cause of microvascular dysfunction. Angiotensin II was indeed found to be implicated in the pathogenesis of obesity-associated hypertension and insulin resistance, possibly through interference with the vascular effects of insulin.

Increased aldosterone levels have also been associated with resistant hypertension and insulin resistance, which is illustrated in patients with primary aldosteronism. Furthermore, aldosterone is known to exert several detrimental effects on the vasculature, some of which are offset by mineralocorticoid receptor antagonists.

In obese individuals, plasma aldosterone concentrations are increased as well. We hypothesize that increased aldosterone levels in adipose persons induce microvascular dysfunction, which contributes to the development of insulin resistance and hypertension, and mineralocorticoid receptor antagonism results in improved insulin sensitivity and decreased blood pressure by counteracting the adverse effects of aldosterone on the microvasculature.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 years
* Caucasian
* Waist circumference > 102 cm (men)/> 88 cm (women)
* Triglycerides > 1.7 mmol/L
* High-normal blood pressure (office blood pressure: 130/85 - 139/89 mm Hg) or stage I hypertension (office blood pressure: 140/90 mm Hg - 159/99 mm Hg; 24h ABPM: 125/80 - 149/89 mm Hg)

Exclusion Criteria:

* Cardiovascular disease (stroke, coronary artery disease, peripheral vascular disease, congestive heart failure, cardiac shunts, cardiac surgery, pulmonary hypertension, cardiac arrhythmias, family history of cardiac arrhythmias or sudden cardiac death)
* Diabetes mellitus/impaired glucose metabolism (fasting glucose values > 5.6 mmol/L)
* Grade 2 or 3 hypertension (office blood pressure: > 160/100 mm Hg; ABPM > 150/90 mm Hg)
* Unstable or severe pulmonary disease
* Unstable or severe thyroid disorders
* Inflammatory diseases
* Alcohol use > 2 U/day (women)/> 3 U/day (men)
* Use of antihypertensive, lipid-lowering or glucose-lowering medications,
* Use of corticosteroids, medication known to inhibit or induce CYP3A4, lithium, and tricyclic antidepressants or antipsychotic medication, and regular use (weekly or several times a week) of NSAIDs
* Plasma potassium levels < 3.2 mmol/L or > 5 mmol/L
* eGFR < 60 mL/min
* Impairment of hepatic function
* Pregnancy or lactation

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Change in capillary recruitment (insulin-induced increase in microvascular blood volume in skeletal muscle) from baseline after 4 weeks of Eplerenone treatment or placebo | Change from baseline after 4 weeks of treatment with either Eplerenone or placebo
  The difference in microvascular blood volume in skeletal muscle of the forearm, which is assessed with contrast enhanced ultrasound, before and during a hyperinsulinemic, euglycemic clamp (performed to determine insulin sensitivity)

CONTACTS AND LOCATIONS:
Overall Officials: prof. C.D.A. Stehouwer, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands